CLINICAL TRIAL: NCT04934527
Title: Evaluating a Therapeutic Association Between CMV-specific Immunoglobulin Infusion and Pre-transplant CD16-expressing Gamma Delta Vdelta 2 Negative T-cells in CMV-positive Patients for Preventive Treatment of CMV Infection in Renal Transplantation
Brief Title: Association of T Gamma Delta-CD16+ Cells and Anti-CMV Immunoglobulins in the Prevention of CMV Infection
Acronym: SYNTAGME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2020/26
Record Dates: First submitted 2021-04-16; First posted 2021-06-22 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplantation; CMV Infection
Keywords: kidney transplantation; CMV Infection; Tgamma-delta Vdelta2 negativ lymphocyte; Cytotect
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with positive CMV serology at transplantation will receive 6 infusions of Cytotect every 15 days with the first injection on the day of transplantation. CMV infection will be monitored by quantitative PCR on whole blood every week during 3 months and then every 2 weeks until 4 months and then at months 5 and 6, 9 and 12.
  Interventions: Drug: Cytotect

INTERVENTIONS:
Drug: Cytotect — The inclusion visit is conducted by the investigating nephrologist and the patient will receive their first infusion of anti-CMV Ig.
  Patients with positive CMV serology at transplantation will receive 6 infusions of 100 units per kilogram of body weight every 15 days with the first injection on the day of transplantation, i.e. at visits D0, S2, S4, S6, S8 and S10. CMV infection will be monitored by quantitative PCR on whole blood every week during 3 months and then every 2 weeks until 4 months and then at months 5 and 6, 9 and 12.

SUMMARY:
CMV infection in transplantation remains the most frequent infectious complication causing increased morbidity and mortality. International recommendations advocate prevention of this infection by instituting direct antiviral treatment or monitoring viral replication by PCR with the start of curative antiviral treatment when the DNAemia is positive.

The risk of CMV infection varies according to the serostatus of the donor (D) and recipient (R) at the time of transplantation. In the absence of prophylaxis, CMV infection occurs in 60-80% of D+R-, 50-60% of D+R+ and 25-50% of D-R+.

The humoral anti-CMV response is represented by the production of antibodies to envelope proteins (gB and gH) and to molecules involved in viral attachment and entry into target cells. However, the majority of CMV-specific antibodies do not have antiviral neutralising activity. The investigators have identified a new player in the specific anti-CMV response expressing the Fc RIIIa receptor (CD16), that interacts with anti-CMV immunoglobulins (Ig): the Tgamma-delta V delta 2-negative lymphocyte (LTgdVd2neg). This lymphocyte subpopulation shows persistent expansion in the peripheral blood of kidney transplant patients with CMV infection. These cells express an effector-memory phenotype (CD45RA+/CD27-). This expansion is associated with resolution of infection in patients. The investigators have shown that CD16 is specifically and constitutively expressed on the surface of CMV-induced LTgdVd2neg in healthy volunteers and kidney transplant patients. The investigators have observed that one of the antiviral activities of anti-CMV IgG lies in its binding to the Fc RIIIa receptor (CD16) on the surface of LTgdVd2neg. The anti-CMV IgGs capturing virions thus activate CD16+ LTgdVd2neg with production of IFN interferon which in turn is responsible for inhibition of CMV viral multiplication.

Anti-CMV IgG is a recommended therapeutic option, with a marketing authorisation for the prevention of CMV infection in kidney transplantation in Europe and a Temporary Authorisation for Use in France.

Thus, R+ patients expressing a significant level of LTgdVd2neg CD16+ at D0 of transplantation could be protected against CMV, in the absence of direct antiviral treatment by the addition of anti-CMV Ig.

DETAILED DESCRIPTION:
SYNTAGME is a single-centre prospective phase II pilot study. Transplant candidates from our centre who meet the inclusion criteria without exclusion criteria will be offered this study. Anti-CMV Ig infusions will be performed the day of transplantation at 100 units per kilo of body weight and then every 15 days for a total of 6 infusions.

Systematic and frequent monitoring for the occurrence of CMV DNAemia will be performed throughout this study. Real-time quantitative CMV PCR on whole blood (WHO standard provided by the National Institute for Biological Standards and Control) will be performed every week until M3, then every fortnight until 4 months and then at months 5, 6, 9 and 12. CMV infection will be defined by the presence of a positive CMV PCR in whole blood. Universal prophylaxis with VALGANCICLOVIR will be prohibited.

Pre-emptive antiviral treatment will be initiated in case of CMV infection, if the DNAemia reaches the threshold chosen by the centre, which is 5000 IU/ml. The choice of treatment will be left to the discretion of the clinician: IV ganciclovir (5mg/Kg/12H) or valganciclovir (900mg/12H) until viral replication is negated. Doses will be adjusted for kidney function using the Cockcroft-Gault formula, in accordance with laboratory recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years of age,
2. Patient candidate for a first transplant or a re-transplantation, registered on the national waiting list of the Biomedicine Agency.
3. CMV seropositive patients (positive serology at pre-transplant assessment or at D0 of transplantation)
4. Patients receiving a kidney transplant from a deceased or living donor.
5. Women of childbearing age with a negative pregnancy test at inclusion and agreeing to the use of effective contraception throughout the study period and two months after the end of the follow-up period.
6. Patient affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

1. CMV negative (R-) patients.
2. Historical or current Graft Incompatible Rate (GIR) > 85%.
3. Patients who have received anti-CMV therapy within 28 days prior to transplantation.
4. Indication for induction therapy with anti-lymphocyte globulin, rituximab, polyvalent intravenous immunoglobulin or any other immunomodulatory molecule, and mTOR inhibitor therapy, which have been described to be associated with a decreased incidence of CMV infection
5. Patients who have received or are receiving a solid organ transplant other than a kidney transplant.
6. Patients known to be seropositive for human immunodeficiency virus (HIV), hepatitis B virus (HBV; HbS Ag positive) or hepatitis C virus (HCV; HCV antibody positive),
7. Known allergy, contraindication or intolerance to specific anti-HCV Ig, mycophenolic acid, basiliximab, corticosteroids, cyclosporine A, tacrolimus or to excipients of these products.
8. Any form of substance abuse, psychiatric disorder or condition that, in the opinion of the investigator, may complicate communication during follow-up.
9. Foreseeable inability to comply with planned protocol visits/reviews.
10. Patients under guardianship/guardianship
11. Pregnant or breastfeeding woman
12. Patients with a contraindication to receiving Cytotect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of CMV infection in the year following transplantation. | 12 months after inclusion day
  Occurrence of CMV infection will assess thanks to LT gdVd2 level 12 months after inclusion day.

SECONDARY OUTCOMES:
Measure the absence of CMV infection in the year following transplantation. | 12 months after inclusion day
  Determining an LTgdCD16+ predictive threshold of an effective therapeutic response to anti-CMV Ig in R+ patients undergoing preventive therapy for post-transplant CMV infection. Thanks to LTgdCD16+ immunophenotyping
Determined the percentage of NK cells in peripheral blood expressing CD16, which may be associated with protection from CMV infection after anti-CMV Ig infusion. | 12 months after inclusion day
  Thanks to NK cells immunophenotyping and CMV PCR
Assessing kinetics of LTgds and NK cells in patients receiving Ig-anti CMV. | 12 months after inclusion day
  Described phenotypic kinetics of LTgds and NK cells, thanks to NK cells and LTgds immunophenotyping.
Assessing the incidence of CMV infection occurring in the first year post-transplant in R+ patients on pre-emptive follow-up receiving CMV Ig. | 12 months after inclusion day
  This outcome will be evaluated by comparing between CMV infection occurring in the first year post-transplant in R+ patients on pre-emptive follow-up receiving CMV Ig and an historical group of R+ patients on the same pre-emptive follow-up but not receiving CMV Ig.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France